CLINICAL TRIAL: NCT01110811
Title: A Randomized Controlled Trial Comparing Transoral Incisionless Fundoplication (TIF) Using EsophyX With Sham Procedure for the Treatment of PPI Dependent GERD: the TIF vs. Sham Study
Brief Title: Transoral Incisionless Fundoplication (TIF) Versus Sham for Treatment of Gastroesophageal Reflux Disease (GERD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EndoGastric Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D2009-10
Record Dates: First submitted 2010-04-23; First posted 2010-04-27 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Gastroesophageal Reflux Disease; Hiatal Hernia
Keywords: GERD; Esophagitis; Fundoplication; Anti-reflux surgery; PPI dependent
MeSH Terms: conditions — Gastroesophageal Reflux; Hernia, Hiatal; Esophagitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- TIF procedure (Active Comparator): Transoral Incisionless Fundoplication (TIF)
  Interventions: Procedure: Transoral Incisionless Fundoplication (TIF)
- Sham procedure (Sham Comparator): The intervention on the Sham procedure consisted of an upper gastrointestinal endoscopy, or EGD.(esophagogastricduodenoscopy).
  Interventions: Procedure: Transoral Incisionless Fundoplication (TIF)

INTERVENTIONS:
Procedure: Transoral Incisionless Fundoplication (TIF) — The TIF procedure results in the creation of an esophago-gastric fundoplication extending up to 4 cm above the Z-line and 270 degress around the esophagus.

SUMMARY:
The study objective is to evaluate the relative merits, safety and effectiveness of transoral incisionless fundoplication (TIF) in proton pump inhibitor (PPI) dependent GERD patients compared with sham procedure.

DETAILED DESCRIPTION:
Primary Effectiveness Endpoint: The proportion of patients in clinical remission after 6 months (without being classified as treatment failure).

Secondary Effectiveness: PPI consumption, esophageal acid exposure, reduction in QOLRAD and GSRS scores and healing of reflux esophagitis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* On daily PPIs for > 6 months
* Documented PPI dependency
* Persistent GERD symptoms without PPI therapy during the titration phase of the study
* Evidence of two or more of the following while off PPI therapy (> 10 days):
* Erosive esophagitis (Los Angeles grade A-C)
* Abnormal ambulatory pH study
* Moderate to severe GERD symptoms
* Normal or near normal esophageal motility (by manometry)
* Patient willing to cooperate with post-operative dietary recommendations and assessment tests
* Signed informed consent

Exclusion Criteria:

* BMI > 35
* Hiatal hernia > 3 cm
* Esophagitis LA grade D
* Esophageal ulcer
* Esophageal stricture
* Barretts esophagus (Prague: C>1, M>2)
* Esophageal motility disorder
* Severe gastric paralysis
* Pregnancy or plans for pregnancy in the next 12 months
* Immunosuppression
* ASA > 2
* Portal hypertension and/or varices
* History of previous resective gastric or esophageal surgery, cervical spine fusion, Zenker's diverticulum, esophageal epiphrenic diverticulum, achalasia, scleroderma or dermatomyositis, eosinophilic esophagitis, or cirrhosis
* Active gastro-duodenal ulcer disease
* Gastric outlet obstruction or stenosis
* Severe gastroparesis or delayed gastric emptying confirmed by solid-phase gastric emptying study if patient complains of postprandial satiety during assessment
* Coagulation disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-04; Primary Completion 2015-09 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Proportion of patients in clinical remission | at 6 month follow-up
  Fifty nine per cent of patients remained in clinical remission

SECONDARY OUTCOMES:
Reduction in symptoms | at 6 moths follow-up
  GSRS score improved from 14 (range 10-21) to 10 (range 6-19) with P = 0.004.
Normalized esophageal acid exposure | at 6 months follow-up
  Sixty nine per cent of patients (69%) in TIF surgical arm normalized esophageal acid exposure.
Healed reflux esophagitis | at 6 months follow-up
  In 80% of patients healing of esophagitis was observed

CONTACTS AND LOCATIONS:
Overall Officials: Lars Lundell, M.D., Principal Investigator — Karolinska University, Huddinge Hospital, Stockholm, Sweden
Locations (4):
- University Hospitals Leuven, Leuven, Belgium
- University of Nantes Hospital, Nantes, France
- Sweden (2):
  - Karolinska University, Ersta Hospital, Stockholm
  - Karolinska University, Huddinge Hospital, Stockholm

REFERENCES:
- [Derived] Hakansson B, Montgomery M, Cadiere GB, Rajan A, Bruley des Varannes S, Lerhun M, Coron E, Tack J, Bischops R, Thorell A, Arnelo U, Lundell L. Randomised clinical trial: transoral incisionless fundoplication vs. sham intervention to control chronic GERD. Aliment Pharmacol Ther. 2015 Dec;42(11-12):1261-70. doi: 10.1111/apt.13427. Epub 2015 Oct 13. PMID 26463242